CLINICAL TRIAL: NCT02124902
Title: A Co-clinical Trial in Triple Negative Breast Cancer Patients With Genoproteomic Discovery
Brief Title: Neoadjuvant Treatment of Triple Negative Breast Cancer Patients With Docetaxel and Carboplatin to Assess Anti-tumor Activity
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient funding/staff
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); Breast Cancer Research Foundation (Other); NeoImmuneTech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201404107; 1U24CA209837-01A1 (NIH)
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Results first posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-10

CONDITIONS: Triple Negative Breast Neoplasms
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Washington University: Neoadjuvant docetaxel and carboplatin (Experimental): Docetaxel will be administered intravenously at a dose of 75mg/m2 over 60 minutes on Day 1 of each 21-day cycle. Carboplatin AUC 6 will be administered intravenously over 30 minutes on Day 1 of each 21-day cycle immediately following docetaxel infusion. A total of 6 cycles will be given.
  Interventions: Drug: Docetaxel; Drug: Carboplatin; Procedure: FDG-PET/MR
- Baylor: Neoadjuvant docetaxel and carboplatin (Experimental): Docetaxel will be administered intravenously at a dose of 75mg/m2 over 60 minutes on Day 1 of each 21-day cycle. Carboplatin AUC 6 will be administered intravenously over 30 minutes on Day 1 of each 21-day cycle immediately following docetaxel infusion.
  Interventions: Drug: Docetaxel; Drug: Carboplatin; Procedure: FDG-PET/MR

INTERVENTIONS:
Drug: Docetaxel
  Other Names: Docefrez®, Taxotere®
Drug: Carboplatin
  Other Names: Paraplatin, Paraplatin-AQ
Procedure: FDG-PET/MR — * Prior to initialization of Cycle 1 and completion of cycle 1 (preferably on cycle 2 day 1)
  * This is not optional for final 30 participants enrolled on the study

SUMMARY:
This is a single arm open label phase II study in women with clinical stage 2 or 3 triple negative breast cancer to assess the anti-tumor activity (in terms of pathologic complete response rate) of neoadjuvant docetaxel in combination with carboplatin. Patient derived xenografts will also be developed simultaneously for the purposes of genoproteomic analysis.

Please note that Baylor College of Medicine (BCM) has a parallel study the same as this study. Baylor is expected to enroll approximately 19 participants that have complied with the inclusion and exclusion criteria for this study (excluded participants from BCM will include male participants or participants with inflammatory breast cancer). The investigators will pool participants and data from the BCM study and the study at Washington University School of Medicine. Pooling the data will potentially improve statistical power.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed AJCC7 clinical stage II or III breast cancer with complete surgical excision of the breast cancer after neoadjuvant chemotherapy as the treatment goal.
* Patients with PR+ tumors are allowed.
* HER2 negative by FISH or IHC staining 0 or 1+.
* ER less than Allred score of 3 or less than 1% positive staining cells in the invasive component of the tumor
* Tumor size at least 2cm in one dimension by clinical or radiographic exam (WHO criteria). Patients with palpable lymph nodes may be enrolled regardless of tumor size.
* At least 18 years of age.
* ECOG performance status ≤ 2
* Normal bone marrow and organ function as defined below:

  * Leukocytes ≥ 3,000/mcL
  * Absolute neutrophil count ≥ 1,500/mcl
  * Platelets ≥ 100,000/mcl
  * Serum bilirubin within (or under ) normal limits (OR total bilirubin ≤ 3.0 x IULN with direct bilirubin within normal range in patients with well documented Gilbert Syndrome)
  * AST(SGOT)/ALT(SGPT) within (or under ) normal limits
  * Creatinine clearance ≥ 60 mL/min/1.73 m2
* Patients may be pre- or post-menopausal. Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).
* Able to tolerate PET/MRI with intravenous contrast administration and must complete the applicable MRI screening evaluation form

Exclusion Criteria:

* Prior systemic therapy for the indexed breast cancer.
* A history of other malignancy ≤ 5 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix.
* Patients with bilateral or inflammatory breast cancer.
* Currently receiving any other investigational agents.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to docetaxel or carboplatin.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding. Patient must have a negative serum pregnancy test within 7 days of study entry if premenopausal.
* Known HIV-positivity.
* Sentinel lymph node biopsy
* Renal insufficiency (glomerular filtration rate (GFR) < 30 mL/min/1.73 m2) measured within the past 60 days which precludes safe administration of the contrast agent
* On dialysis
* Prior allergic reaction to gadolinium-based MR contrast agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2014-07-07 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Foluso Ademuyiwa, M.D., MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ademuyiwa FO, Chen I, Luo J, Rimawi MF, Hagemann IS, Fisk B, Jeffers G, Skidmore ZL, Basu A, Richters M, Ma CX, Weilbaecher K, Davis J, Suresh R, Peterson LL, Bose R, Bagegni N, Rigden CE, Frith A, Rearden TP, Hernandez-Aya LF, Roshal A, Clifton K, Opyrchal M, Akintola-Ogunremi O, Lee BH, Ferrando-Martinez S, Church SE, Anurag M, Ellis MJ, Gao F, Gillanders W, Griffith OL, Griffith M. Immunogenomic profiling and pathological response results from a clinical trial of docetaxel and carboplatin in triple-negative breast cancer. Breast Cancer Res Treat. 2021 Aug;189(1):187-202. doi: 10.1007/s10549-021-06307-3. Epub 2021 Jun 26. PMID 34173924
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Washington University: Neoadjuvant Docetaxel and Carboplatin: Docetaxel will be administered intravenously at a dose of 75mg/m^2 over 60 minutes on Day 1 of each 21-day cycle. Carboplatin AUC 6 will be administered intravenously over 30 minutes on Day 1 of each 21-day cycle immediately following docetaxel infusion. A total of 6 cycles will be given.
- Baylor: Neoadjuvant Docetaxel and Carboplatin: Docetaxel will be administered intravenously at a dose of 75mg/m^2 over 60 minutes on Day 1 of each 21-day cycle. Carboplatin AUC 6 will be administered intravenously over 30 minutes on Day 1 of each 21-day cycle immediately following docetaxel infusion.
Period: Overall Study
Arm/Group | Washington University: Neoadjuvant Docetaxel and Carboplatin | Baylor: Neoadjuvant Docetaxel and Carboplatin
Started (Completion is considered receiving 6 cycles of treatment.) | 123 | 25
Completed | 106 | 19
Not Completed | 17 | 6
Not completed — Adverse Event | 7 | 2
Not completed — Went to alternative treatment | 4 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Not eligible | 1 | 0
Not completed — Did not receive carboplatin in cycle 6 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Washington University: Neoadjuvant Docetaxel and Carboplatin | Baylor: Neoadjuvant Docetaxel and Carboplatin | Total
Number analyzed (Participants) | 123 | 25 | 148
Age, Continuous [Median (Full Range); unit: years] | 53 [25 to 77] | 57 [29 to 71] | 53 [25 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 25 | 148
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 9 | 9
  Not Hispanic or Latino | 123 | 16 | 139
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 32 | 1 | 33
  White | 89 | 22 | 111
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 123 | 25 | 148

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response (pCR) Rate
Description: -A patient is considered to not to have a pCR if any of the following are true:
  * There is histologic evidence of invasive tumor cells in the surgical breast specimen or the axillary lymph nodes.
  * The patient has discontinued neoadjuvant treatment early due to refusal, toxicity, or radiographic evidence of progression and then goes straight to surgery where there is histologic evidence of invasive tumor cells in the surgical breast specimen and the axillary lymph nodes
  * The patient has discontinued neoadjuvant treatment early due to refusal, toxicity or radiographic evidence of progression and then receives alternative treatment.
  * The patient discontinues study treatment, refuses surgery, or is unable to undergo surgery due to a co-morbid condition.
  Thus, any patient who does not receive alternative treatment prior to surgery and has no histologic evidence of invasive tumor cells in the surgical breast specimen and the axillary lymph nodes is considered to have a pCR.
Time Frame: At the time of surgery (surgery will take place 3-5 weeks after completion of treatment and estimated treatment length is 18 weeks)
Population: 17 participants from Washington University were not evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Washington University: Neoadjuvant Docetaxel and Carboplatin | Baylor: Neoadjuvant Docetaxel and Carboplatin
Number analyzed (Participants) | 106 | 25
Participants | 47 | 11

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment through 30 days after completion of treatment. Treatment could continue for a total of 6 cycles and each cycle is 21 days in length. All-cause mortality was followed from start of treatment through completion of follow-up. Follow-up for survival is for 5 years.
Arm/Group | Washington University: Neoadjuvant Docetaxel and Carboplatin | Baylor: Neoadjuvant Docetaxel and Carboplatin
All-Cause Mortality (participants affected / at risk) | 9/123 | 3/25
Serious Adverse Events (participants affected / at risk) | 21/123 | 3/25
Other Adverse Events (participants affected / at risk) | 123/123 | 16/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Washington University: Neoadjuvant Docetaxel and Carboplatin (N=123) | Baylor: Neoadjuvant Docetaxel and Carboplatin (N=25)
Anemia (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 0
Diverticulitis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Oral thrush (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Fever (General disorders) | 1 | 0
Pain (General disorders) | 2 | 0
Pain in extremity (General disorders) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Rash pustular (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Neutrophil count decreased (Investigations) | 3 | 0
Platelet count decreased (Investigations) | 2 | 0
White blood cell decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Protein calorie malnutrition (Metabolism and nutrition disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Acute cystitis without gross hematuria (Renal and urinary disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 2 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Washington University: Neoadjuvant Docetaxel and Carboplatin (N=123) | Baylor: Neoadjuvant Docetaxel and Carboplatin (N=25)
Anemia (Blood and lymphatic system disorders) | 108 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Non-cardiac chest pain (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 4 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 4 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 0
Blurred vision (Eye disorders) | 3 | 0
Dacryostenosis (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 5 | 0
Epiphora (Eye disorders) | 1 | 0
Eye stye (Eye disorders) | 3 | 0
Eye twitching (Eye disorders) | 3 | 0
Itchy eyes (Eye disorders) | 1 | 0
Viral conjunctivitis (Eye disorders) | 1 | 0
Watering eyes (Eye disorders) | 18 | 0
Abdominal pain (Gastrointestinal disorders) | 14 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0
Bloating (Gastrointestinal disorders) | 2 | 0
Blood in stool (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 2 | 0
Colonic fistula (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 64 | 0
Diarrhea (Gastrointestinal disorders) | 63 | 4
Diverticulitis (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0
Dysgeusia (Gastrointestinal disorders) | 4 | 0
Dyspepsia (Gastrointestinal disorders) | 45 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Esophageal spasms (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 6 | 0
Mucositis oral (Gastrointestinal disorders) | 48 | 1
Nausea (Gastrointestinal disorders) | 81 | 0
Oral dysesthesia (Gastrointestinal disorders) | 2 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Stomach pain (Gastrointestinal disorders) | 2 | 0
Tender gums (Gastrointestinal disorders) | 1 | 0
Thrush (Gastrointestinal disorders) | 5 | 0
Toothache (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 48 | 1
Back pain (General disorders) | 1 | 0
Boil pain (General disorders) | 1 | 0
Chills (General disorders) | 16 | 0
Cramps (General disorders) | 2 | 0
Edema face (General disorders) | 3 | 0
Edema limbs (General disorders) | 37 | 0
Edema trunk (General disorders) | 1 | 0
Fatigue (General disorders) | 95 | 1
Fever (General disorders) | 12 | 0
Knee pain (General disorders) | 1 | 0
Localized edema (General disorders) | 2 | 0
Malaise (General disorders) | 1 | 0
Mild body aches (General disorders) | 1 | 0
Neck edema (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 7 | 0
Overall pain & muscle spasms (General disorders) | 1 | 0
Pain (General disorders) | 26 | 0
Tongue numbness (General disorders) | 1 | 0
Whole body pain (General disorders) | 1 | 0
Anorectal infection (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0
Cold (Infections and infestations) | 2 | 0
Cold sore (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Eye infection (Infections and infestations) | 2 | 0
Food poisoning (Infections and infestations) | 1 | 0
Head cold (Infections and infestations) | 1 | 0
Herpes, left thigh (Infections and infestations) | 1 | 0
Infection: Yeast and gums (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Mucosal infection (Infections and infestations) | 1 | 0
Papulopustular rash (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Pink eye (Infections and infestations) | 1 | 0
Possible cellulitis at port site (Infections and infestations) | 1 | 0
Shingles (Infections and infestations) | 3 | 0
Sinusitis (Infections and infestations) | 2 | 0
Skin infection (Infections and infestations) | 2 | 2
Staph infection (secondary to spider bite) (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Upper respiratory infection (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 18 | 0
Urinary tract infection symptoms (Infections and infestations) | 1 | 0
Vaginal infection (Infections and infestations) | 7 | 0
Wound infection (Infections and infestations) | 2 | 0
Yeast infection (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0
Bruising (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 28 | 0
Alkaline phosphatase increased (Investigations) | 5 | 0
Aspartate aminotransferase increased (Investigations) | 9 | 0
Blood bilirubin increased (Investigations) | 3 | 0
Creatinine increased (Investigations) | 8 | 0
INR increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 68 | 2
Neutrophil count decreased (Investigations) | 27 | 2
Platelet count decreased (Investigations) | 82 | 2
Weight gain (Investigations) | 3 | 0
Weight loss (Investigations) | 11 | 0
White blood cell decreased (Investigations) | 36 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 60 | 1
Dehydration (Metabolism and nutrition disorders) | 10 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 11 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 26 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 3 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 13 | 0
Hypochoremia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 15 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 7 | 1
Hyponatremia (Metabolism and nutrition disorders) | 16 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 17 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 | 0
Left hip pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 25 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 40 | 0
Dysgeusia (Nervous system disorders) | 53 | 0
Headache (Nervous system disorders) | 44 | 0
Lightheadedness (Nervous system disorders) | 3 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 2 | 0
Peripheral motor neuropathy (Nervous system disorders) | 5 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 75 | 2
Presyncope (Nervous system disorders) | 3 | 0
Sciatic nerve (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 4 | 0
Tremor (Nervous system disorders) | 1 | 0
Vasovagal reaction (Nervous system disorders) | 1 | 0
Vasovagal syncope (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 9 | 0
Depression (Psychiatric disorders) | 12 | 0
Insomnia (Psychiatric disorders) | 33 | 0
Restlessness (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 2 | 0
Hematuria (Renal and urinary disorders) | 2 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 2 | 0
Dyspareunia (Reproductive system and breast disorders) | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0
Vaginal dryness (Reproductive system and breast disorders) | 2 | 0
Vaginal pain (Reproductive system and breast disorders) | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 26 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 50 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oral sensitivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Runny nose (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus drainage with dry cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 101 | 0
Brittle nails (Skin and subcutaneous tissue disorders) | 2 | 0
Bug sting on thumb (Skin and subcutaneous tissue disorders) | 1 | 0
Diffuse itchy rash (bug bites) (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 18 | 0
Dry, cracked hands (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Finger nail pain (Skin and subcutaneous tissue disorders) | 3 | 0
Folliculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 23 | 0
Hypohidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Moles and freckles (Skin and subcutaneous tissue disorders) | 1 | 0
Mouth crack (Skin and subcutaneous tissue disorders) | 2 | 0
Nail bed changes (Skin and subcutaneous tissue disorders) | 2 | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | 31 | 0
Nail loss (Skin and subcutaneous tissue disorders) | 6 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 5 | 0
Nail tenderness (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 7 | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Rash (NOS) (Skin and subcutaneous tissue disorders) | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 11 | 0
Redness on skin of feet (Skin and subcutaneous tissue disorders) | 1 | 0
Scalp pain (Skin and subcutaneous tissue disorders) | 2 | 0
Skin burn on knuckles (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 | 0
Skin peeling (Skin and subcutaneous tissue disorders) | 4 | 0
Tender nails (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 4 | 0
Hot flashes (Vascular disorders) | 31 | 0
Hypertension (Vascular disorders) | 42 | 0
Hypotension (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/02/NCT02124902/Prot_SAP_000.pdf